CLINICAL TRIAL: NCT03534557
Title: FEV1/FEV6 and FEV6 as an Alternative for FEV1/FVC and FVC in the Detection of Airway Obstruction in a Small Group of Bolivian Subjects
Brief Title: FEV1/FEV6 and FEV6 as an Alternative for FEV1/FVC and FVC in Bolivian Subjects
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Giuseppe Liistro, Head of clinic, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: StLucFEV6
Record Dates: First submitted 2018-05-08; First posted 2018-05-23 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Copd
Keywords: spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD: FEV1/FVC and FEV1/FEV6 will be compared within the same cohort of COPD patients
  Interventions: Diagnostic Test: FEV6 spirometry

INTERVENTIONS:
Diagnostic Test: FEV6 spirometry — During the same spirometry, to compare the relative value of FVC and FEV6

SUMMARY:
Comparison of FEV1/FEV6 and FEV6 as an alternative for FEV1/FVC and FCV in the detection of airway obstruction in a Bolivian population

DETAILED DESCRIPTION:
The data of consecutive adult smoker patients, referred to the Clínica del Pulmón (Santa Cruz, Bolivia), between May 2018 and June 2018, will be analyzed. All the patients are current or ex-smokers, complaining of dyspnea, cough or expectorations. Spirometry measurements will be performed with a Medisoft Body Box 5500 by one highly trained and experienced pulmonologist according to the guidelines of the ATS/ERS.

The criteria used to detect airway obstruction are either the fixed cut-off points according to GOLD recommendations (FEV1/FVC<0.70) or the lower limit of normal (FEV1/FVC<LLN). These indices will be compared to a fixed cut-off FEV1/FEV6 <0.73 as proposed by Vandevoorde et al. or to a FEV1/FV6 ration < LLN. Reference equations used are those of Caucasians from the NHANES III survey.

Statistical tests will be done using IBM SPSS 24 software. Cohen's κ will be used to determine if there is an agreement between the definitions of airway obstruction.

ELIGIBILITY:
Inclusion Criteria:

* adult smoker suspected of COPD

Exclusion Criteria:

* unable to perform spirometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
The aim of this preliminary study is to determine if the criteria of airway obstruction using FEV6 as a surrogate of FVC are transposable to a non-selected Bolivian population | one measurement lasts 10 minutes
  see above

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Liistro, MD,PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Clínica del Pulmón, Santa Cruz, Bolivia

IPD SHARING:
Plan to Share IPD: Undecided